CLINICAL TRIAL: NCT07083011
Title: A Three-Arm, Observational, Pilot Study of 68Ga-Fibroblast Activation Protein Inhibitor (FAPI) Positron Emission Tomography in Heart Failure
Brief Title: A Study of 68Ga-Fibroblast Activation Protein Inhibitor (FAPI) Positron Emission Tomography in Heart Failure
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Omar Abou Ezzeddine, Principal Investigator, Mayo Clinic
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: 25-004043
Record Dates: First submitted 2025-07-16; First posted 2025-07-24 (Actual); Last update posted 2025-09-25 (Actual); Status verified 2025-09

CONDITIONS: Heart Failure With Preserved Ejection Fraction
MeSH Terms: interventions — 68Ga-FAPI

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (3):
- Obese subjects with HFpEF (heart failure with preserved ejection fraction) (Experimental)
  Interventions: Drug: 68Ga-FAPI (gallium-68-labeled fibroblast activation protein inhibitor)
- Active cardiac sarcoidosis (Active Comparator)
  Interventions: Drug: 68Ga-FAPI (gallium-68-labeled fibroblast activation protein inhibitor)
- Healthy subjects (Active Comparator)
  Interventions: Drug: 68Ga-FAPI (gallium-68-labeled fibroblast activation protein inhibitor)

INTERVENTIONS:
Drug: 68Ga-FAPI (gallium-68-labeled fibroblast activation protein inhibitor) — 68Ga-FAPI is a gallium-68 fibroblast activation protein inhibitor that will be injected into subjects during a PET (positron emission tomography) scan

SUMMARY:
The purpose of this study is to assess the performance of 68Ga- FAPI PET in heart failure with preserved ejection fraction (HFpEF)

ELIGIBILITY:
HFpEF Group Inclusion:

* Patients aged ≥ 30 years old with exertional dyspnea (NYHA II and III) and LVEF ≥50%
* BMI ≥ 30
* New diagnosis of HFpEF based on RHC at baseline (elevated PCWP at rest and/or during exercise)

HFpEF Group Exclusion:

* Primary cardiomyopathy or pericardial disease or ≥ moderate valvular disease
* Dyspnea due to lung disease or CAD
* Severe anemia, liver, or renal disease
* Active cancer
* Systemic active inflammatory or autoimmune disease (e.g. rheumatoid arthritis, SLE, etc.)
* Recent hospitalization (< 30 days) or coronary revascularization (< 90 days)
* Patients already taking SGLT2i and/or GLP-1A
* Pregnant or breastfeeding
* Inability to tolerate supine position for the PET/CT or CMR scans.
* Contraindications for safe CMR scanning (e.g., uncontrolled claustrophobia, cochlear implant, implanted neural stimulator)
* Known gadolinium allergy
* Presence of implantable cardiac pacemaker or defibrillator or mechanical valve.

Cardiac Sarcoid Group Inclusion:

* Ambulatory patients aged ≥ 18 years old
* New referrals to the Sarcoid Clinic with a confirmed but untreated diagnosis of definite or probable CS based on 2014 HRS consensus (see Table 2)
* With a positive cardiac 18F-FDG PET scan within 30 days.

Cardiac Sarcoid Group Exclusion:

* Already on immunosuppressive therapy
* Pregnant or breastfeeding
* Severe liver or renal disease (estimated GFR < 30 or dialysis-dependent)
* Recent coronary revascularization (< 90 days)
* Active cancer
* Known gadolinium allergy
* Inability to tolerate supine position for the PET/CT or CMR scans.
* Contraindications for safe CMR scanning (e.g., uncontrolled claustrophobia, cochlear implant, implanted neural stimulator)
* Presence of implantable cardiac pacemaker or defibrillator or mechanical valve.

Healthy Controls Group Inclusion:

* Adults ≥ 30 years old
* No major chronic disease (cardiopulmonary, inflammatory, autoimmune, cancer, renal or liver impairment, etc.)
* No intake of relevant medication, defined as regular intake of at least one of the following: anticoagulants, antiplatelets, antihypertensive / diuretics, antidiabetics, antiarrhythmic, immunosuppressants, chemotherapy, antibiotics/antivirals/antifungals

Healthy Controls Group Exclusion:

* BMI ≥ 30
* Pregnant or breastfeeding
* Known gadolinium allergy
* Inability to tolerate supine position for the PET/CT or CMR scans.
* Contraindications for safe CMR scanning (e.g., uncontrolled claustrophobia, cochlear implant, implanted neural stimulator)

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 35 (Estimated)
Dates: Start 2025-11 (Estimated); Primary Completion 2027-07 (Estimated); Study Completion 2027-07 (Estimated)

PRIMARY OUTCOMES:
Myocardial 68Ga-FAPI (68Ga-Fibroblast Activation Protein Inhibitor) volume | Baseline and 6 Months
  Myocardial 68Ga-FAPI volume will be determined by a PET (positron emission tomography) scan and measured in cm3
Mean Standardized Uptake Value (SUVmean) and Max Standardized Uptake Value (SUVmax) | Baseline and 6 Months
  SUVmean and SUVmax will be determined by a PET (positron emission tomography) scan and measured as a dimensionless ratio
Area of 68Ga-FAPI (68Ga-Fibroblast Activation Protein Inhibitor) uptake | Baseline and 6 Months
  Area of 68Ga-FAPI will be determined by a PET (positron emission tomography) scan and measured as a % of polar map.
68Ga-FAPI target-to-background ratio | Baseline and 6 Months
  68Ga-FAPI target-to-background ratio will be determined by a PET (positron emission tomography) scan and measured as a dimensionless ratio.

CONTACTS AND LOCATIONS:
Overall Officials: Omar Abou Ezzeddine, M.D, M.S, Principal Investigator — Mayo Clinic; Gregorio Tersalvi, M.D, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic in Rochester, Rochester, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No